CLINICAL TRIAL: NCT01030289
Title: The Effectiveness of tDCS in Decreasing Food Cravings
Brief Title: The Effectiveness of Transcranial Direct Current Stimulation (tDCS) in Decreasing Food Cravings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Jeffrey Borckardt, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Borckardt_19429
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Craving
Keywords: food cravings

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- real tDCS First Visit (Active Comparator): On the First Visit, A single 20-minute tDCS session will be conducted using 2.0mA current. Using the international 10-20 EEG system, the anode will be placed over F4, which corresponds to the right dorsolateral prefrontal cortex (DLPFC), and the cathode will be placed over F3, which corresponds to the left dorsolateral prefrontal cortex. Electrodes will be standard sponge electrodes soaked In a sterile solution of .9% sodium chloride insulated by a latex casing.
  Interventions: Device: real tDCS
- sham tDCS First Visit (Sham Comparator): On the First Visit, For sham tDCS, the device will be turned on for 30 seconds and then turned off for the duration of the 20-minute session.
  Interventions: Device: sham tDCS
- real tDCS Second Visit (Active Comparator): Participant returns for the second visit 48-72 hours after completing the first visit. A single 20-minute tDCS session will be conducted using 2.0mA current. Using the international 10-20 EEG system, the anode will be placed over F4, which corresponds to the right dorsolateral prefrontal cortex (DLPFC), and the cathode will be placed over F3, which corresponds to the left dorsolateral prefrontal cortex. Electrodes will be standard sponge electrodes soaked In a sterile solution of .9% sodium chloride insulated by a latex casing.
  Interventions: Device: real tDCS
- sham tDCS Second Visit (Sham Comparator): Participant returns for the second visit 48-72 hours after completing the first visit. For sham tDCS, the device will be turned on for 30 seconds and then turned off for the duration of the 20-minute session.
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: real tDCS — transcranial direct current stimulation
  Arms: real tDCS First Visit; real tDCS Second Visit
Device: sham tDCS — transcranial direct current stimulation
  Arms: sham tDCS First Visit; sham tDCS Second Visit

SUMMARY:
This study aims to evaluate the effectiveness of transcranial direct current stimulation (tDCS) in decreasing food cravings. Specifically, this study will determine whether healthy subjects will report decreased food craving following a single 20-minute session of tDCS (compared to sham tDCS) delivered during and immediately following the exposure to food stimuli.

DETAILED DESCRIPTION:
Recently, the use of low amplitude direct current stimulation of the human cortex has received attention as a possible for treatment for depression and pain (Been et al, 2007). This technique (called transcranial direct current stimulation or tDCS) involves the placement of two sponge electrodes over separate areas of the scalp. tDCS has been shown to be capable of changing the excitability of the superficial neurons immediately beneath the sponge electrodes. Evidence suggests that anodal stimulation is associated with increased cortical excitability and cathodal stimulation is associated with decreased cortical excitability (Been et al, 2007).

Brain imaging studies are beginning to elucidate the functional neuroanatomy of cravings (George, Anton, Bloomer, Teneback, Drobes, Lorberbaum, et al., 2001; Myrick, Anton, Li, Henderson, Drobes, Voronin, et al., 2004). While the role of the prefrontal cortex in regulating cravings remains somewhat unclear, frontal cortical areas appear to be involved in integrating incoming sensory information (such as sights, smells, and sounds) with affective/emotional information in the brain, and may be involved in regulating emotional reactions to various stimuli (Alexander, DeLong, & Strick, 1986; Lorenz, Minoshima, & Casey, 2003). The dorsal lateral prefrontal cortex may become activated when an individual is presented with cues that trigger reward memories associated with certain consumptive behaviors (Anton, 1999). One fMRI study found that when alcoholic subjects were presented with alcohol related cues, there was greater activation in the left prefrontal cortex and anterior thalamus, compared to when they viewed non-alcohol cues (George et al., 2001). Other studies on bulimia and drug cravings have identified hyperactivity in the orbitofrontal cortex and anterior cingulate cortex associated with increases in cravings ratings (Goldstein & Volkow, 2002; Uher, et al., 2004).

Very few studies have attempted to directly manipulate activation of brain structures that might be involved in cravings. tDCS allows researchers to selectively activate or inhibit different brain structures that might play a role in craving behaviors. Previous research with manipulating the activation of brain structures found that alcohol cravings decreased among individuals with alcohol dependence who received either left or right anodal stimulation of the dorsolateral prefrontal cortex (Boggio et al., 2008). This finding, combined with prior functional neuroanatomical work, and research on the relation of food cravings and nicotine cravings suggesting they share a common biologic mechanism (Pepino, Finkbiener, Menella 2009, 2007), suggests that the prefrontal cortex may be a reasonable preliminary tDCS cortical target for potentially inhibiting food cravings.

To date, there has only been one published study examining the relationship between tDCS and food craving. Fregni and colleagues (2008) found cravings to be reduced by anode right/cathode left tDCS and cravings did not increase after anode left/cathode right tDCS. The evidence on the effectiveness of tDCS for decreasing food craving indicates relatively short-lived effects (lasting only a few weeks). While this may ultimately limit the utility of tDCS, it may have a place in the prevention and management of obesity.

This study aims to evaluate the effectiveness of transcranial direct current stimulation (tDCS) in decreasing food cravings. Specifically, this study will determine whether healthy subjects will report decreased food craving following a single 20-minute session of tDCS (compared to sham tDCS) delivered during and immediately following the exposure to food stimuli.

ELIGIBILITY:
Inclusion Criteria:

* 21-70 years of age

Exclusion Criteria:

* pregnant
* history of seizures or epilepsy
* family history or seizures
* history of eating disorder
* history of depression
* taking medications that have been shown to lower seizure threshold
* metal implanted above the waist
* history of autoimmune or endocrine disorders
* diabetes
* allergy to latex
* allergy to peanuts
* brain tumors or lesions

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Goldman, MA, Principal Investigator — Medical University of South Carolina
Locations (1):
- Brain Stimulation Laboratory, Institute of Psychiatry, Charleston, South Carolina, United States

REFERENCES:
- [Background] Goldman RL, Borckardt JJ, Frohman HA, O'Neil PM, Madan A, Campbell LK, Budak A, George MS. Prefrontal cortex transcranial direct current stimulation (tDCS) temporarily reduces food cravings and increases the self-reported ability to resist food in adults with frequent food craving. Appetite. 2011 Jun;56(3):741-6. doi: 10.1016/j.appet.2011.02.013. Epub 2011 Feb 23. PMID 21352881
- See also: Link to Published Results — http://www.ncbi.nlm.nih.gov/pubmed/21352881

RESULTS

PARTICIPANT FLOW:
Groups:
- Real tDCS: On the First Visit, A single 20-minute tDCS session will be conducted using 2.0mA current. Using the international 10-20 EEG system, the anode will be placed over F4, which corresponds to the right dorsolateral prefrontal cortex (DLPFC), and the cathode will be placed over F3, which corresponds to the left dorsolateral prefrontal cortex. Electrodes will be standard sponge electrodes soaked In a sterile solution of .9% sodium chloride insulated by a latex casing.
  Participant returns for the second visit 48-72 hours after completing the first visit to receive real tDCS.
- Sham tDCS: On the First Visit, For sham tDCS, the device will be turned on for 30 seconds and then turned off for the duration of the 20-minute session.
  Participant returns for the second visit 48-72 hours after completing the first visit to receive another session of sham tDCS.
Period: Overall Study
Arm/Group | Real tDCS | Sham tDCS
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 19 met all inclusion/exclusion criteria and completed both study sessions.
Groups:
- All Study Participants: All participants enrolled in the study
Arm/Group | All Study Participants
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.47 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Food Cravings
Description: Twenty-four images of food were presented in random order using a custom developed computer program. While viewing the food images, participants used a computerized visual analog scale to rate how much they would like to eat each food right now if it were actually available to them, how much they liked the food, and how much would they be able to resist tasting the food if it were in front of them. They viewed the pictures and rated before treatment and after real tDCS and Sham tDCS. The scale ranged from 0 (no food cravings) to 100 (extreme food cravings).
  The before treatment after treatment food craving ratings were used to calculate percent change.
Time Frame: before treatment, after treatment
Measure: Mean (Standard Deviation); unit: percentage of change in cravings
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 9 | 10
percentage of change in cravings | -26.81 (26.11) | -7.8 (41.87)

2. Secondary Outcome: Cravings for Sweet Foods
Description: Twenty-four images of food were presented in random order using a custom developed computer program. While viewing the food images, participants used a computerized visual analog scale to rate how much they would like to eat each food right now if it were actually available to them, how much they liked the food, and how much would they be able to resist tasting the food if it were in front of them. They viewed the pictures and rated before treatment and after real tDCS and Sham tDCS. The scale ranged from 0 (no sweet food cravings) to 100 (extreme sweet food cravings).
  The before treatment after treatment ratings for sweet food craving were used to calculate percent change.
Time Frame: before treatment, after treatment
Measure: Mean (Standard Deviation); unit: percentage of change in cravings
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 9 | 10
percentage of change in cravings | -30.5 (23.03) | -0.95 (59.85)

3. Secondary Outcome: Cravings for Carbohydrate Foods
Description: Twenty-four images of food were presented in random order using a custom developed computer program. While viewing the food images, participants used a computerized visual analog scale to rate how much they would like to eat each food right now if it were actually available to them, how much they liked the food, and how much would they be able to resist tasting the food if it were in front of them. They viewed the pictures and rated before treatment, during, and after real tDCS and Sham tDCS. The scale ranged from 0 (no food cravings) to 100 (extreme food cravings).
  The before treatment, during treatment, and after treatment ratings for carbohydrates were used to calculate percent change.
Time Frame: before treatment, during treatment, after treatment
Measure: Mean (Standard Deviation); unit: percentage of change in cravings
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 9 | 10
percentage of change in cravings
  before treatment to during treatment | -24.41 (41.67) | 22.10 (79.12)
  before treatment to after treatment | -25.45 (45.6) | 14.87 (70.12)

4. Secondary Outcome: Inability to Resist Food and tDCS Condition
Description: Twenty-four images of food were presented in random order using a custom developed computer program. While viewing the food images, participants used a computerized visual analog scale to rate how much they would like to eat each food right now if it were actually available to them, how much they liked the food, and how much would they be able to resist tasting the food if it were in front of them. They viewed the pictures and rated before, during, and after real tDCS and Sham tDCS. The scale ranged from 0 (no food cravings, completely resist food) to 100 (extreme food cravings, unable to resist food).
  The before treatment, during treatment, and after treatment resist ratings for carbohydrates were used to calculate percent change.
Time Frame: before treatment, during treatment, after treatment
Measure: Mean (Standard Deviation); unit: percentage of change in resist ratings
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 9 | 10
percentage of change in resist ratings
  before treatment to during treatment | 26.79 (33.71) | 10.66 (39.57)
  before treatment to after treatment | 30.36 (30.82) | 13.38 (39.52)

5. Secondary Outcome: Food Ingested and tDCS Condition
Description: Food was presented on a plate for the participants to eat after treatment. Each participant received a Chocolate Plate, Donut Plate, Cookie Plate, and a Potatoe Chip Plate. Each participant received the same amount of food on each plate. Each plate was weighed in grams separately before and after eating the food. A difference score was calculated to determine how much food was eaten for each type of food.
  The mean difference score was calculated for each type of food for the Sham tDCS group & the Real tDCS group. The means and standard deviations of percent change in the decrease of food (weighed in grams) ingested post-tDCS treatment are reported below for the real tDCS group and the sham tDCS group.
Time Frame: After treatment
Measure: Mean (Standard Deviation); unit: percent change in grams of food ingested
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 9 | 10
percent change in grams of food ingested
  Chocolate | 2.7 (2.8) | 3.9 (6.4)
  Cookies | 7.3 (12.7) | 7.2 (11.6)
  Potato Chips | 6.7 (9.1) | 11.2 (14.0)
  Donuts | 9.1 (16.8) | 7.0 (11.5)

6. Secondary Outcome: Confidence Ratings in Guessing of Treatment Condition
Description: At the end of the participants' second appointment, they were asked to guess which tDCS session was real and which was sham. 0=completely guessing. 10=absolutely sure. We calculated how many participants correctly guessed when they received real and when they received sham. A composite index was created to control for correct-guessing in the mixed model analysis. A new variable was created wherein the "guess correct" value (0=incorrect guess, 1=correct guess) was multiplied by the guess confidence rating for each participant. Thus, those that guess incorrectly had a guess-composite value of 0 whereas those that guessed correctly had a value equal to their guess confidence.
Time Frame: After treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Subjects: All 19 Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 19
units on a scale | 6.45 (2.7)

ADVERSE EVENTS:
Time Frame: 3 days
Groups:
- Real tDCS; Sham tDCS: transcranial direct current stimulation: transcranial direct current stimulation
Arm/Group | Real tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No